CLINICAL TRIAL: NCT05167877
Title: Studying Aging, Mobility and Chronic Low Back Pain in Older Adults Using Remote Monitoring
Brief Title: Aging, Mobility and Chronic Low Back Pain
Status: Active, not recruiting | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Other Study IDs: 21-011
Record Dates: First submitted 2021-11-15; First posted 2021-12-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain; Chronic Pain
Keywords: Low Back Pain; Chronic; Older Adults; Mobility; Remote Monitoring
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Participants without CLBP. Measurements include: bio-physiological, neurophysiological measurements at baseline. Remote monitoring of gait, physical activity for 7 days using inertial measurement unit (IMU) with wearable devices.
  Interventions: Other: No intervention will be given to the participants
- Active group: Participants with CLBP. Measurements include: bio-physiological, neurophysiological measurements at baseline. Remote monitoring of gait, physical activity for 7 days using inertial measurement unit (IMU) with wearable devices. Self-reported measures of pain and type of activity for 7 days using electronic dairy.
  Interventions: Other: No intervention will be given to the participants

INTERVENTIONS:
Other: No intervention will be given to the participants — This is an observational feasibility study with no intervention.

SUMMARY:
Chronic low back pain (CLBP) is very common in older adults and is one of the most common reasons for disability and poor quality of life. Lack of physical activity is considered to negatively impact CLBP and show an inverse association with pain symptoms and limitations.

Remote and real-time monitoring can allow ecological momentary assessment which involves repeated sampling of participants' current behaviors and experiences in their natural environments. Recent advances allow monitoring of activity using inertial measurement units (consisting of accelerometers, gyroscopes and magnetometers) that can be worn by an individual at home or during work.

In our study, we plan to test the feasibility and acceptability of the wearable devices in elderly patients with CLBP and to explore the use of data analytics and machine learning on the recorded data, in order to demonstrate the feasibility of a larger cohort study.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a common condition in elderly population. CLBP is associated with disability and poor quality of life worldwide. Studies have found that the lack of physical activity may negatively impact CLBP and show an inverse association with pain symptoms and limitations. For example, a study demonstrates that physically active patients with CLBP experience less pain [- 0.6, 95% confidence interval (CI): - 1.0 to - 0.1; 0-10 numerical pain scale] and disability (- 8.7, 95% CI: - 14.2 to - 3.1; 0-100 disability scale) compared to patients not adequately active. However, most reports are based on younger adults or using cross-sectional studies with no continuous or real-life monitoring.

Functionally, pain with movement is more important than resting pain. This is especially true of CLBP, which increases in severity with movement. Physical activity has health benefits, including for chronic pain conditions. However, many pain patients suffer from kinesiophobia and consider exercise to be unhelpful. There is uncertainty around exercise induced analgesia, as well as the type of activity in musculoskeletal pain. The present approach to pain recording, suffers from limitations including recall, and does not relate to associated physical activity. With this, the primary drivers of pain-sensory, psychological, and motor factors are studied in isolation. Additionally, objective markers of analgesia and neuroplasticity related to physical activity have not been well studied. There is a paradoxical relationship between physical activity to treat pain and participation in physical activity evoking pain. Most studies on movement evoked pain have been using paradigms of experimental movements which are not natural to patients, and do not consider the influence of contextual factors. Remote and real-time monitoring provides us possibility of measuring the subjects' real-time behaviors and experience. The wearable remote devices are developed to monitor activity and provide large data for various analyses.

The investigators will use an inertial measurement unit (IMU)-based device containing accelerometer, gyroscope and magnetometer worn on each ankle (like a watch) in the current study. The device is capable of measuring spatiotemporal gait parameters (such as asymmetry, variability, speed, stride time, stance to swing ratio, minimum foot clearance) along with type and amount of physical activity. The investigators will capture real-time pain intensity, type, and context of activity using an electronic diary in the form of a wristwatch. Data from both devices will be integrated for processing and analysis, including the use of machine learning and data analytics to develop predictive models. In the present proposal (the first phase), the investigators will use these devices on older adults with mobility (>65 years and <80 years) with (active group) or without CLBP (control group). In this phase, the investigators plan to complete the feasibility and acceptability of these devices and obtain pilot data to support the applications for the larger study funding. After the first phase, the investigators plan to conduct a larger cohort study in older adult CLBP patients using the study devices and applications at the participants' home/living settings.

ELIGIBILITY:
Inclusion Criteria:

* Age >65 and <80 years
* patients with present and known history of non-specific chronic low back pain (CLBP) will be included in the active group
* participants without CLBP will be included in the control group
* ability to comprehend or understand commands in English language

Exclusion Criteria:

* Presence of any unstable cardio-respiratory comorbidity such as congestive heart failure, severe coronary disease, severe chronic obstructive pulmonary disease, or asthma needing daily treatment with puffers
* known history of neurocognitive impairment
* known history of untreated or uncontrolled psychological disorders
* history of previous back surgery
* presence of moderate to severe knee, ankle, or foot pain, and other physical impairments needing walking assistance
* participants expected to receive a new medication treatment or injection for their CLBP during the study week

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly patients without chronic low back pain (CLBP) for control group, and elderly patients with CLBP for active group.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Total time and patterns of wearing the study devices | 7 days
  To assess the compliance of the wearable devices (MetaMotionS IMU to be worn on both of a participant's ankles), time and patterns (all the time, part of the time and when) of wearing them during the study period will be measured with consistent data capture by the devices.
System Usability Scale (SUS) (ranges from 0 to 100; a higher score indicates better acceptability) | On Day 7
  At the end of study, the SUS questionnaire will used to assess participants' acceptability of wearing of the study devices.

SECONDARY OUTCOMES:
Back Performance Scale (BPS) (range from 0 to 15; a higher score indicates worse performance) | At baseline
  The association between BPS measured at baseline and chronic low back pain will be assessed.
Self-paced walking test | At baseline
  Distance (unit: metres) completed in the self-paced two-minute walk test will be measured at baseline. The association between this value and chronic low back pain will be assessed.
Neurophysiological markers | At baseline
  The association between the neurophysiological markers measured from transcranial magnetic stimulation at baseline and chronic low back pain will be assessed.
Gait and physical activity | 7 days
  The association between the physical activity measured using remote monitoring during the study period and chronic low back pain will be assessed.
Subgroups of chronic low back pain (CLBP) | 7 days
  All the collected data including the baseline variables and parameters measured with activity monitoring will be used to explore subgroups of CLBP using effective machine learning methods.

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Shanthanna, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Souza IMB, Sakaguchi TF, Yuan SLK, Matsutani LA, do Espirito-Santo AS, Pereira CAB, Marques AP. Prevalence of low back pain in the elderly population: a systematic review. Clinics (Sao Paulo). 2019 Oct 28;74:e789. doi: 10.6061/clinics/2019/e789. eCollection 2019. PMID 31664424
- [Result] Wong AYL, Karppinen J, Samartzis D. Low back pain in older adults: risk factors, management options and future directions. Scoliosis Spinal Disord. 2017 Apr 18;12:14. doi: 10.1186/s13013-017-0121-3. eCollection 2017. PMID 28435906
- [Result] Deyo RA, Weinstein JN. Low back pain. N Engl J Med. 2001 Feb 1;344(5):363-70. doi: 10.1056/NEJM200102013440508. No abstract available. PMID 11172169
- [Result] Alsufiany MB, Lohman EB, Daher NS, Gang GR, Shallan AI, Jaber HM. Non-specific chronic low back pain and physical activity: A comparison of postural control and hip muscle isometric strength: A cross-sectional study. Medicine (Baltimore). 2020 Jan;99(5):e18544. doi: 10.1097/MD.0000000000018544. PMID 32000363
- [Result] Pinto RZ, Ferreira PH, Kongsted A, Ferreira ML, Maher CG, Kent P. Self-reported moderate-to-vigorous leisure time physical activity predicts less pain and disability over 12 months in chronic and persistent low back pain. Eur J Pain. 2014 Sep;18(8):1190-8. doi: 10.1002/j.1532-2149.2014.00468.x. Epub 2014 Feb 27. PMID 24577780
- [Result] Amorim AB, Pappas E, Simic M, Ferreira ML, Jennings M, Tiedemann A, Carvalho-E-Silva AP, Caputo E, Kongsted A, Ferreira PH. Integrating Mobile-health, health coaching, and physical activity to reduce the burden of chronic low back pain trial (IMPACT): a pilot randomised controlled trial. BMC Musculoskelet Disord. 2019 Feb 11;20(1):71. doi: 10.1186/s12891-019-2454-y. PMID 30744606
- [Result] Corbett DB, Simon CB, Manini TM, George SZ, Riley JL 3rd, Fillingim RB. Movement-evoked pain: transforming the way we understand and measure pain. Pain. 2019 Apr;160(4):757-761. doi: 10.1097/j.pain.0000000000001431. No abstract available. PMID 30371555
- [Result] Hodges PW, Smeets RJ. Interaction between pain, movement, and physical activity: short-term benefits, long-term consequences, and targets for treatment. Clin J Pain. 2015 Feb;31(2):97-107. doi: 10.1097/AJP.0000000000000098. PMID 24709625
- [Result] Kosek E, Roos EM, Ageberg E, Nilsdotter A. Increased pain sensitivity but normal function of exercise induced analgesia in hip and knee osteoarthritis--treatment effects of neuromuscular exercise and total joint replacement. Osteoarthritis Cartilage. 2013 Sep;21(9):1299-307. doi: 10.1016/j.joca.2013.06.019. PMID 23973144
- [Result] Thomas KS, Muir KR, Doherty M, Jones AC, O'Reilly SC, Bassey EJ. Home based exercise programme for knee pain and knee osteoarthritis: randomised controlled trial. BMJ. 2002 Oct 5;325(7367):752. doi: 10.1136/bmj.325.7367.752. PMID 12364304
- [Result] Vincent HK, Seay AN, Montero C, Conrad BP, Hurley RW, Vincent KR. Kinesiophobia and fear-avoidance beliefs in overweight older adults with chronic low-back pain: relationship to walking endurance--part II. Am J Phys Med Rehabil. 2013 May;92(5):439-45. doi: 10.1097/PHM.0b013e318287633c. PMID 23478452
- [Result] Holden MA, Nicholls EE, Young J, Hay EM, Foster NE. Role of exercise for knee pain: what do older adults in the community think? Arthritis Care Res (Hoboken). 2012 Oct;64(10):1554-64. doi: 10.1002/acr.21700. PMID 22511582
- [Result] Nijs J, Kosek E, Van Oosterwijck J, Meeus M. Dysfunctional endogenous analgesia during exercise in patients with chronic pain: to exercise or not to exercise? Pain Physician. 2012 Jul;15(3 Suppl):ES205-13. PMID 22786458
- [Result] Hurwitz EL, Morgenstern H, Chiao C. Effects of recreational physical activity and back exercises on low back pain and psychological distress: findings from the UCLA Low Back Pain Study. Am J Public Health. 2005 Oct;95(10):1817-24. doi: 10.2105/AJPH.2004.052993. PMID 16186460
- [Result] Hoffman SL, Johnson MB, Zou D, Harris-Hayes M, Van Dillen LR. Effect of classification-specific treatment on lumbopelvic motion during hip rotation in people with low back pain. Man Ther. 2011 Aug;16(4):344-50. doi: 10.1016/j.math.2010.12.007. Epub 2011 Jan 20. PMID 21256073
- [Result] Butera KA, Fox EJ, George SZ. Toward a Transformed Understanding: From Pain and Movement to Pain With Movement. Phys Ther. 2016 Oct;96(10):1503-1507. doi: 10.2522/ptj.20160211. No abstract available. PMID 27694519
- [Result] Thibaut A, Zeng D, Caumo W, Liu J, Fregni F. Corticospinal excitability as a biomarker of myofascial pain syndrome. Pain Rep. 2017 Apr 18;2(3):e594. doi: 10.1097/PR9.0000000000000594. eCollection 2017 May. PMID 29392210
- [Result] Chaves AR, Snow NJ, Alcock LR, Ploughman M. Probing the Brain-Body Connection Using Transcranial Magnetic Stimulation (TMS): Validating a Promising Tool to Provide Biomarkers of Neuroplasticity and Central Nervous System Function. Brain Sci. 2021 Mar 17;11(3):384. doi: 10.3390/brainsci11030384. PMID 33803028
- [Result] Knell G, Gabriel KP, Businelle MS, Shuval K, Wetter DW, Kendzor DE. Ecological Momentary Assessment of Physical Activity: Validation Study. J Med Internet Res. 2017 Jul 18;19(7):e253. doi: 10.2196/jmir.7602. PMID 28720556
- [Result] Majumder S, Mondal T, Deen MJ. A Simple, Low-Cost and Efficient Gait Analyzer for Wearable Healthcare Applications. IEEE Sensors Journal. 2019;19(6):2320-2329.
- [Result] Jin B, Thu TH, Baek E, Sakong S, Xiao J, Mondal T, Deen MJ. Walking-age analyzer for healthcare applications. IEEE J Biomed Health Inform. 2014 May;18(3):1034-42. doi: 10.1109/JBHI.2013.2296873. PMID 24808231
- [Result] Bennett MI, Smith BH, Torrance N, Potter J. The S-LANSS score for identifying pain of predominantly neuropathic origin: validation for use in clinical and postal research. J Pain. 2005 Mar;6(3):149-58. doi: 10.1016/j.jpain.2004.11.007. PMID 15772908
- [Result] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, Delitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. Phys Ther. 2015 Feb;95(2):e1-e18. doi: 10.2522/ptj.2015.95.2.e1. PMID 25639530
- [Result] Huang W, Rose AJ, Bayliss E, Baseman L, Butcher E, Garcia RE, Edelen MO. Adapting summary scores for the PROMIS-29 v2.0 for use among older adults with multiple chronic conditions. Qual Life Res. 2019 Jan;28(1):199-210. doi: 10.1007/s11136-018-1988-z. Epub 2018 Sep 12. PMID 30209722
- [Result] Deyo RA, Katrina Ramsey, Buckley DI, Michaels L, Kobus A, Eckstrom E, Forro V, Morris C. Performance of a Patient Reported Outcomes Measurement Information System (PROMIS) Short Form in Older Adults with Chronic Musculoskeletal Pain. Pain Med. 2016 Feb;17(2):314-24. doi: 10.1093/pm/pnv046. PMID 26814279
- [Result] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Result] Davidson M, Keating JL. A comparison of five low back disability questionnaires: reliability and responsiveness. Phys Ther. 2002 Jan;82(1):8-24. doi: 10.1093/ptj/82.1.8. PMID 11784274
- [Result] Strand LI, Moe-Nilssen R, Ljunggren AE. Back Performance Scale for the assessment of mobility-related activities in people with back pain. Phys Ther. 2002 Dec;82(12):1213-23. PMID 12444880
- [Result] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Result] Kim E, Lovera J, Schaben L, Melara J, Bourdette D, Whitham R. Novel method for measurement of fatigue in multiple sclerosis: Real-Time Digital Fatigue Score. J Rehabil Res Dev. 2010;47(5):477-84. doi: 10.1682/jrrd.2009.09.0151. PMID 20803391
- [Result] Keogh A, Dorn JF, Walsh L, Calvo F, Caulfield B. Comparing the Usability and Acceptability of Wearable Sensors Among Older Irish Adults in a Real-World Context: Observational Study. JMIR Mhealth Uhealth. 2020 Apr 20;8(4):e15704. doi: 10.2196/15704. PMID 32310149